CLINICAL TRIAL: NCT01884519
Title: Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix/Influsplit SSW 2013/2014 in People 18 Years of Age and Above
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Influenza Vaccine, Fluarix®/Influsplit SSW® (2013/2014 Season), in Adults 18 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200160; 2013-000855-42 (EudraCT Number)
Record Dates: First submitted 2013-06-13; First posted 2013-06-24 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: Elderly; Influenza; Safety; Adults; Immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- Fluarix/Influsplit 18-60 Years Group (Experimental): Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: Fluarix/Influsplit SSW® (2013-2014 season)
- Fluarix/Influsplit > 60 Years Group (Experimental): Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
  Interventions: Biological: Fluarix/Influsplit SSW® (2013-2014 season)

INTERVENTIONS:
Biological: Fluarix/Influsplit SSW® (2013-2014 season) — 1 dose administered intramuscularly (or deeply subcutaneously) in the deltoid region of the non-dominant arm

SUMMARY:
The purpose of this study is to assess, in adults 18 years of age and above, the immunogenicity and reactogenicity of the seasonal influenza vaccine, Fluarix/Influsplit SSW 2013/2014, containing the three vaccine influenza strains (two A strains and one B strain) for the 2013/2014 season.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female aged 18 years or above at the time of vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or subjects with well-controlled chronic diseases as established by medical history and clinical examination before entering the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of vaccination.

Exclusion Criteria:

* Participation in previous year's Fluarix registration study (116663).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within the six months prior to vaccination. Inhaled and topical steroids are allowed.
* Any administration of a long-acting immune-modifying drug within 6 months before study start, or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned administration during the study period.
* Administration of an influenza vaccine within the twelve months preceding the study vaccination.
* Receipt of a vaccine other than the study vaccine within 30 days before study vaccination and/or plan to receive any vaccine other than the study vaccine during the entire study period.
* Clinically or virologically confirmed influenza infection within the six months preceding the study vaccination.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C/99.5°F on oral, axillary or tympanic setting, or ≥ 38.0°C/100.4°F on rectal setting. The preferred route for recording temperature in this study will be axillary.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Acute, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic underlying disease (such as cancer, chronic obstructive pulmonary disease under oxygen therapy, insulin-dependent diabetes mellitus), not stabilized or clinically serious.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of Guillain-Barré syndrome.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine including latex.
* Anaphylaxis following the administration of vaccine(s).
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study or would make intramuscular injection unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-07-01; Primary Completion 2013-08-02 (Actual); Study Completion 2013-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Germany (4):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (11.5) | 68.2 (5.49) | 55.4 (15.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Vaccine Influenza Strains
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 0 and Day 21
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Titer
  H1N1, Day 0 | 27.3 [20.3 to 36.8] | 15.7 [12.1 to 20.4]
  H1N1, Day 21 | 444.6 [335.6 to 588.9] | 197.0 [142.6 to 272.1]
  H3N2, Day 0 | 15.8 [11.9 to 21.1] | 14.2 [11.0 to 18.4]
  H3N2, Day 21 | 73.8 [57.8 to 94.2] | 80.0 [58.4 to 109.5]
  Yamagata, Day 0 | 105.0 [83.6 to 131.8] | 95.2 [77.5 to 116.9]
  Yamagata, Day 21 | 424.6 [347.6 to 518.8] | 327.5 [266.2 to 402.9]

2. Primary Outcome: Number of Subjects Who Were Seroprotected for Anti-HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  H1N1, Day 0 | 25 | 14
  H1N1, Day 21 | 58 | 56
  H3N2, Day 0 | 12 | 12
  H3N2, Day 21 | 50 | 44
  Yamagata, Day 0 | 53 | 55
  Yamagata, Day 21 | 60 | 60

3. Primary Outcome: Number of Seroconverted Subjects for Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroconverted subjects was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  H1N1 | 44 | 46
  H3N2 | 31 | 29
  Yamagata | 30 | 23

4. Primary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Fold increase
  H1N1 | 16.3 [10.8 to 24.5] | 12.6 [8.7 to 18.2]
  H3N2 | 4.7 [3.4 to 6.4] | 5.6 [4.0 to 7.9]
  Yamagata | 4.0 [3.1 to 5.3] | 3.4 [2.7 to 4.3]

5. Primary Outcome: Number of Subjects With Seroprotection Power (SPP) for HI Antibody Titer Against Each of the Three Vaccine Influenza Strains Above the Cut-off Value.
Description: SPP was defined as the number of vaccinated subjects with a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:40. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 48 | 48
Subjects
  H1N1 [N=35,46] | 33 | 42
  H3N2 [N=48,48] | 38 | 32
  Yamagata [N=7,5] | 7 | 5

6. Secondary Outcome: Humoral Immune Response in Terms of HI Antibody Titers Against Each of the Three Vaccine Influenza Strains
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2 influenza seasons prior to season 2012/2013.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Fluarix/Influsplit 18-60 Years Group With Vaccination: Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0 and who had received an influenza vaccine during the 2 influenza seasonal prior to season 2012-2013. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluarix/Influsplit 18-60 Years Group Without Vaccination: Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0 and who had not received an influenza vaccine during the 2 influenza seasonal prior to season 2012-2013. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluarix/Influsplit > 60 Years Group With Vaccination: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0 and who had received an influenza vaccine during the 2 influenza seasonal prior to season 2012-2013. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluarix/Influsplit > 60 Years Group Without Vaccination: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0 and who had not received an influenza vaccine during the 2 influenza seasonal prior to season 2012-2013. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluarix/Influsplit 18-60 Years Group With Vaccination | Fluarix/Influsplit 18-60 Years Group Without Vaccination | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 20 | 40 | 29 | 31
Titers
  H1N1, Day 0 | 28.7 [17.2 to 48.1] | 26.6 [18.2 to 38.9] | 16.3 [10.5 to 25.2] | 15.1 [10.9 to 21.0]
  H1N1, Day 21 | 348.8 [200.3 to 607.4] | 501.9 [361.0 to 698.0] | 158.2 [99.1 to 252.5] | 241.9 [152.7 to 383.3]
  H3N2, Day 0 | 18.6 [10.8 to 32.0] | 14.6 [10.3 to 20.8] | 17.3 [11.4 to 26.2] | 11.8 [8.6 to 16.2]
  H3N2, Day 21 | 60.6 [39.3 to 93.5] | 81.4 [60.0 to 110.4] | 58.6 [39.9 to 86.2] | 106.9 [65.6 to 174.3]
  Yamagata, Day 0 | 109.3 [74.3 to 160.9] | 102.9 [76.7 to 138.0] | 110.6 [84.6 to 144.5] | 82.7 [60.3 to 113.4]
  Yamagata, Day 21 | 355.0 [247.3 to 509.5] | 464.4 [362.9 to 594.2] | 237.3 [184.2 to 305.8] | 442.6 [328.9 to 595.7]

7. Secondary Outcome: Number of Subjects Who Were Seroprotected for Anti-HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2 influenza seasons prior to season 2012/2013.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- Fluarix/Influsplit 18-60 Years Group With Vaccination: Subjects 18-60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluarix/Influsplit 18-60 Years Group Without Vaccination: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluarix/Influsplit 18-60 Years Group With Vaccination | Fluarix/Influsplit 18-60 Years Group Without Vaccination | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 20 | 40 | 29 | 31
Subjects
  H1N1, Day 0 | 9 | 16 | 8 | 6
  H1N1, Day 21 | 19 | 39 | 26 | 30
  H3N2, Day 0 | 5 | 7 | 6 | 6
  H3N2, Day 21 | 16 | 34 | 20 | 24
  Yamagata, Day 0 | 18 | 35 | 29 | 26
  Yamagata, Day 21 | 20 | 40 | 29 | 31

8. Secondary Outcome: Number of Seroconverted Subjects for Anti-HA Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2 influenza seasons prior to season 2012/2013.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group With Vaccination | Fluarix/Influsplit 18-60 Years Group Without Vaccination | Fluarix/Influsplit > 60 Years Group With Vaccination | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 20 | 40 | 29 | 31
Subjects
  H1N1 | 13 | 31 | 20 | 26
  H3N2 | 8 | 23 | 10 | 19
  Yamagata | 6 | 24 | 5 | 18

9. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2 influenza seasons prior to season 2012/2013.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Groups:
- Fluarix/Influsplit > 60 Years Group With Vaccinationars Group: Subjects above 60 years of age received 1 dose of Fluarix/Influsplit SSW 2013-2014 vaccine at Day 0 and who had received an influenza vaccine during the 2 influenza seasonal prior to season 2012-2013. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluarix/Influsplit 18-60 Years Group With Vaccination | Fluarix/Influsplit 18-60 Years Group Without Vaccination | Fluarix/Influsplit > 60 Years Group With Vaccinationars Group | Fluarix/Influsplit > 60 Years Group Without Vaccination
Number analyzed (Participants) | 20 | 40 | 29 | 31
Fold increase
  H1N1 | 12.1 [5.8 to 25.4] | 18.9 [11.4 to 31.4] | 9.7 [5.5 to 17.0] | 16.0 [9.7 to 26.5]
  H3N2 | 3.3 [2.0 to 5.2] | 5.6 [3.7 to 8.3] | 3.4 [2.4 to 4.8] | 9.1 [5.3 to 15.5]
  Yamagata | 3.2 [2.0 to 5.2] | 4.5 [3.2 to 6.3] | 2.1 [1.7 to 2.7] | 5.4 [3.9 to 7.4]

10. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were ecchymosis, induration, pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 ecchymosis, induration, redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any Ecchymosis | 0 | 0
  Grade 3 Ecchymosis | 0 | 0
  Any Induration | 0 | 2
  Grade 3 Induration | 0 | 0
  Any Pain | 38 | 15
  Grade 3 Pain | 0 | 0
  Any Redness | 8 | 3
  Grade 3 Redness | 0 | 0
  Any Swelling | 6 | 2
  Grade 3 Swelling | 0 | 0

11. Secondary Outcome: Duration of Solicited Local Symptoms.
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 38 | 15
Days
  Induration [N=0,2] | 0.0 [0.0 to 0.0] | 1.5 [1.0 to 2.0]
  Pain [N=38, 15] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
  Redness [N=8,3] | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 4.0]
  Swelling [N=6,2] | 1.0 [1.0 to 4.0] | 2.0 [2.0 to 2.0]

12. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, increased sweating and fever [axillary temperature above 37.5 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diarrhea and/or abdominal pain. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature above 39.0°C
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any Arthralgia | 5 | 5
  Grade 3 Arthralgia | 0 | 0
  Related Arthralgia | 4 | 3
  Any Fatigue | 10 | 7
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 6 | 4
  Any Gastrointestinal symptoms | 4 | 1
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 3 | 1
  Any Headache | 10 | 5
  Grade 3 Headache | 2 | 0
  Related Headache | 9 | 5
  Any Myalgia | 14 | 5
  Grade 3 Myalgia | 0 | 0
  Related Myalgia | 12 | 4
  Any Shivering | 4 | 0
  Grade 3 Shivering | 0 | 0
  Related Shivering | 4 | 0
  Any Sweating | 3 | 7
  Grade 3 Sweating | 0 | 0
  Related Sweating | 1 | 4
  Any Fever ≥( 37.5°C) | 0 | 1
  Grade 3 Fever (>39.0°C) | 0 | 0
  Related Fever | 0 | 1

13. Secondary Outcome: Duration of Solicited General Symptoms.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 11
Measure: Median (Full Range); unit: Days
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 14 | 7
Days
  Arthralgia [N=5,5] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 4.0]
  Fatigue [N=10, 7] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0]
  Gastrointestinal symptoms [N=4,1] | 1.0 [1.0 to 1.0] | 3.0 [3.0 to 3.0]
  Headache [N=10,5] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Myalgia [N=14,5] | 1.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Sweating [N=3,7] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 4.0]
  Shivering [N=4,0] | 1.0 [1.0 to 1.0] | 0.0 [0.0 to 0.0]
  Fever (Axillary) [N=0,1] | 0.0 [0.0 to 0.0] | 1.0 [1.0 to 1.0]

14. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any Unsolicted AEs | 5 | 3
  Grade 3 Unsolicted AEs | 0 | 0
  Related Unsolicted AEs | 0 | 1

15. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Days 0-180)
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any SAEs | 0 | 0
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 180; Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period; Unsolicited symptoms: During the 21-day (Day 0-20) post-vaccination period
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 47/60 | 24/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix/Influsplit 18-60 Years Group (N=60) | Fluarix/Influsplit > 60 Years Group (N=60)
Pain (General disorders) | 38 | 15
Redness (General disorders) | 8 | 3
Swelling (General disorders) | 6 | 2
Arthralgia (General disorders) | 5 | 5
Fatigue (General disorders) | 10 | 7
Gastrointestinal symptoms (General disorders) | 4 | 1
Headache (General disorders) | 10 | 5
Myalgia (General disorders) | 14 | 5
Shivering (General disorders) | 4 | 0
Sweating (General disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.